CLINICAL TRIAL: NCT03533582
Title: Pediatric Hepatic Malignancy International Therapeutic Trial (PHITT)
Brief Title: Cisplatin and Combination Chemotherapy in Treating Children and Young Adults With Hepatoblastoma or Liver Cancer After Surgery
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHEP1531; NCI-2017-01910 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AHEP1531 (Other: Children's Oncology Group); AHEP1531 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-08

CONDITIONS: Childhood Hepatocellular Carcinoma; Childhood Malignant Liver Neoplasm; Fibrolamellar Carcinoma; Hepatoblastoma; Hepatocellular Malignant Neoplasm, Not Otherwise Specified
MeSH Terms: conditions — Fibrolamellar hepatocellular carcinoma; Hepatoblastoma | interventions — Specimen Handling; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Doxorubicin; Etoposide; Fluorouracil; dehydroftorafur; Gemcitabine; Irinotecan; Oxaliplatin; Watchful Waiting; Observation; Sorafenib; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Group A1 (WDF) (Active Comparator): Patients undergo observation. Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Other: Patient Observation
- GROUP A2 (NON-WDF) (Experimental): Patients receive cisplatin IV over 6 hours on day 1 following surgery. Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin
- GROUP B1 ARM 4-CDDP (Experimental): Patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 14 days for 4 cycles (2 pre-surgery, 2 post-surgery) in the absence of disease progression or unacceptable toxicity. Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin
- GROUP B1 ARM 6-CDDP (Experimental): Patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 14 days for 6 cycles (2 pre-surgery, 4 post-surgery) in the absence of disease progression or unacceptable toxicity. Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Resection
- GROUP B2 ARM I (Experimental): Patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 14 days for up to 6 total cycles (4 pre-surgery, 2 post-surgery). After cycle 4, patients undergo surgery, then continue with 2 additional cycles of cisplatin. Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Resection
- GROUP B2 ARM II (Experimental): Patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 14 days for up to 6 total cycles. Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin
- GROUP C ARM C5VD (Experimental): Patients receive cisplatin IV over 6 hours on day 1, 5-fluorouracil IV over 1-15 minutes, vincristine sulfate IV over 1 minute on days 1, 8, and 15 and doxorubicin IV over 1-15 minutes on days 1 and 2. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo surgery after cycle 2 or 4. Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Drug: Doxorubicin; Drug: Fluorouracil; Drug: Vincristine Sulfate
- GROUP C ARM CDDP (Experimental): Patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 14 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo surgery after cycle 2 or 4. Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Resection
- GROUP D1 (Experimental): SIOPEL-4 INDUCTION: Patients receive cisplatin IV over 6 hours on days 1, 8, and 15 (for cycles 1 and 2) and days 1 and 8 (for cycle 3) and doxorubicin IV over 1-15 minutes on days 8 and 9 during cycles 1 and 2 and days 1 and 2 during cycle 3. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients with lung complete remission (either with chemotherapy and/or surgery) receive carboplatin IV over 1 hour on day 1 and doxorubicin IV over 1-15 minutes on days 1 and 2. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Drug: Doxorubicin
- GROUP D2 ARM CE (Experimental): SIOPEL-4 IV INDUCTION: Patients receive cisplatin IV over 6 hours on days 1, 8, and 15 (for cycles 1 and 2) and days 1 and 8 (for cycle 3) and doxorubicin IV over 1-15 minutes on days 8 and 9. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  Patients receive carboplatin IV over 1 hour on days 1 and 2, doxorubicin IV over 1-15 minutes on days 1 and 2 during cycles 1, 3 and 5, and carboplatin over 1 hour and etoposide IV over 2 hours on day 1 and 2 of cycles 2, 4 and 6. Treatments repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Drug: Doxorubicin; Drug: Etoposide
- GROUP D2 ARM VI (Experimental): SIOPEL-4 IV INDUCTION: Patients receive cisplatin IV over 6 hours on days 1, 8, and 15 (for cycles 1 and 2) and days 1 and 8 (for cycle 3) and doxorubicin IV over 1-15 minutes on days 8 and 9. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  Patients receive carboplatin IV over 1 hour on days 1 and 2 and doxorubicin IV over 1-15 minutes on days 1 and 2 during cycles 1, 3 and 5. Patients also receive vincristine sulfate IV over 1 minute on days 1 and 8 and irinotecan IV over 90 minutes QD on days 1 to 5 of cycles 2, 4 and 6. Treatments repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Drug: Doxorubicin; Drug: Irinotecan; Drug: Vincristine Sulfate
- GROUP E1 (Active Comparator): Patients undergo observation only. Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Other: Patient Observation
- GROUP E2 (PLADO) (Experimental): Patients receive cisplatin IV over 6 hours on day 1 and doxorubicin IV over 1-15 minutes on days 1 and 2 following surgery. Treatments repeat every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Drug: Doxorubicin
- GROUP F ARM 1 (PLADO) (Experimental): Patients receive cisplatin IV over 6 hours on day 1, doxorubicin IV over 1-15 minutes on days 1 and 2 and sorafenib PO BID on days 3-21. Treatments repeat every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients may undergo surgery, if tumors are resectable, or receive an additional 3 cycles of the treatment. Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Drug: Doxorubicin; Drug: Sorafenib
- GROUP F ARM 2 (P/GEMOX) (Experimental): Patients receive cisplatin IV over 6 hours on day 1, doxorubicin IV over 1-15 minutes on days 1 and 2 and sorafenib PO BID on days 3-14 of cycles 1 and 3. Patients also receive gemcitabine IV over 90 minutes on day 1, oxaliplatin IV over 2 hours on day 1 and sorafenib PO on days 1-14 of cycles 2 and 4. Patients may undergo surgery, if tumors are resectable, or receive an additional 4 cycles of the treatment. Patients may optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Drug: Doxorubicin; Drug: Gemcitabine; Drug: Oxaliplatin; Procedure: Resection; Drug: Sorafenib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: GROUP D1; GROUP D2 ARM CE; GROUP D2 ARM VI
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: GROUP A2 (NON-WDF); GROUP B1 ARM 4-CDDP; GROUP B1 ARM 6-CDDP; GROUP B2 ARM I; GROUP B2 ARM II; GROUP C ARM C5VD; GROUP C ARM CDDP; GROUP D1; GROUP D2 ARM CE; GROUP D2 ARM VI; GROUP E2 (PLADO); GROUP F ARM 1 (PLADO); GROUP F ARM 2 (P/GEMOX)
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
  Arms: GROUP C ARM C5VD; GROUP D1; GROUP D2 ARM CE; GROUP D2 ARM VI; GROUP E2 (PLADO); GROUP F ARM 1 (PLADO); GROUP F ARM 2 (P/GEMOX)
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
  Arms: GROUP D2 ARM CE
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: GROUP C ARM C5VD
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
  Arms: GROUP F ARM 2 (P/GEMOX)
Drug: Irinotecan — Given IV
  Arms: GROUP D2 ARM VI
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; Elplat; JM 83; JM-83; JM83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; RP54780; SR 96669; SR-96669; SR96669
  Arms: GROUP F ARM 2 (P/GEMOX)
Other: Patient Observation — Undergo watchful waiting
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: GROUP E1; Group A1 (WDF)
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection
  Arms: GROUP B1 ARM 6-CDDP; GROUP B2 ARM I; GROUP C ARM CDDP; GROUP F ARM 2 (P/GEMOX)
Drug: Sorafenib — Given PO
  Other Names: BA4 43 9006; BAY 43 9006; BAY 43-9006; BAY 439006; BAY-43-9006; Bay-439006; BAY439006
  Arms: GROUP F ARM 1 (PLADO); GROUP F ARM 2 (P/GEMOX)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: GROUP C ARM C5VD; GROUP D2 ARM VI

SUMMARY:
This partially randomized phase II/III trial studies how well, in combination with surgery, cisplatin and combination chemotherapy works in treating children and young adults with hepatoblastoma or hepatocellular carcinoma. Drugs used in chemotherapy, such as cisplatin, doxorubicin, fluorouracil, vincristine sulfate, carboplatin, etoposide, irinotecan, sorafenib, gemcitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving combination chemotherapy may kill more tumor cells than one type of chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To reduce therapy associated toxicity for patients with non-metastatic hepatoblastoma (HB) and hepatocellular carcinoma (HCC) without adversely affecting long term outcomes.

II. To determine the event-free survival (EFS) in patients with HB whose tumor is completely resected at diagnosis and either receive no adjuvant chemotherapy (completely resected well differentiated fetal [WDF] histology HB) or 2 cycles of standard dose cisplatin monotherapy (completely resected non-well differentiated fetal histology HB - 100 mg/m^2/cycle given 3 weeks apart). (Group A) III. To demonstrate that 4 to 6 cycles of interval compressed lower dose cisplatin monotherapy (80 mg/m^2/cycle; 320-480 mg/m^2 total) is adequate for low risk HB. (Group B) IIIa. In patients who are resected after 2 cycles of cisplatin monotherapy, to compare EFS following a randomized comparison of 2 versus 4 post-operative cycles of cisplatin monotherapy. (Group B) IIIb. In patients whose tumors are deemed unresectable after 2 cycles of cisplatin monotherapy, to determine the proportion of tumors rendered completely resectable by an additional 2 or 4 cycles of chemotherapy. (Group B) IV. To compare in a randomized fashion, EFS in patients with intermediate risk HB treated with 6 cycles of cisplatin/5-fluorouracil/vincristine/doxorubicin (C5VD) chemotherapy versus 6 cycles of interval compressed cisplatin monotherapy (100 mg/m^2/dose). (Group C) V. To determine the EFS in patients with HCC whose tumor is completely resected at diagnosis who receive no adjuvant chemotherapy (completely resected HCC arising in the context of underlying liver disease) or 4 cycles of cisplatin/doxorubicin (PLADO) (completely resected de novo HCC). (Group E) VI. To improve the EFS of patients with high risk HB by treating them with interval compressed cisplatin and doxorubicin based induction regimen followed by response-adapted consolidation therapy. (Group D) VIa. In patients whose metastatic disease resolves with the administration of Societe Internationale d'Oncologie Pediatrique (SIOPEL) 4 Induction therapy, to determine if the promising pilot results observed in SIOPEL 4 can be validated in a large international study. (Group D1) VIb. In patients whose metastatic disease does not resolve with the administration of SIOPEL 4 Induction therapy, to determine in a randomized comparison which post induction treatment (irinotecan and vincristine sulfate [vincristine] alternating with carboplatin and doxorubicin or carboplatin and etoposide alternating with carboplatin and doxorubicin) results in superior outcomes. (Group D Arm CE & Arm VI) VII. In patients with unresectable/metastatic HCC at diagnosis, to determine whether the addition of gemcitabine and oxaliplatin (GEMOX + sorafenib) to a cisplatin, doxorubicin and sorafenib backbone improves chemotherapy response, resectability and survival. (Group F)

EXPLORATORY OBJECTIVES:

I. To determine if the Childhood Hepatic tumor International Consortium (CHIC) hepatoblastoma risk stratification analysis of very low risk (Group A), low risk (Group B), intermediate risk (Group C) and high risk (Group D) groups stratifies patients allowing appropriate utilization of varying intensity chemotherapy regimens and surgical resection strategies.

II. To define the prognostic relevance of a positive microscopic margin in Group A-D resected HB specimens.

III. To define the frequency of histologically detectable multifocal lesions in liver explants and resected specimens in which multifocal disease was detected at diagnosis and disappeared on cross sectional imaging following treatment with chemotherapy.

IV. To define the prognostic relevance in HB of a 'small cell undifferentiated' tumor component and percentage of tumor necrosis in post chemotherapy specimens.

V. To determine the prognostic impact on EFS and overall survival (OS) of biopsy technique in liver tumors unresectable at diagnosis.

VI. To determine the 3-year EFS and OS of HB patients who undergo liver transplantation vs extreme resection in Group C and D patients.

VII. To determine the 3-year EFS and OS of Group D patients who undergo pulmonary metastasectomy.

VIII. To determine the 3-year EFS and OS of patients who undergo liver transplantation for HCC.

IX. To determine the frequency of relapse in non-metastatic HCC in children treated by liver transplantation versus conventional resection.

X. To determine the concordance of Pretreatment Extent of Disease (PRETEXT) and Post-treatment Extent of disease (POSTTEXT) based surgical guidelines and the surgical intervention performed.

XI. To collect for future analysis, HB and HCC tumor specimens that can be molecularly characterized to validate newly identified molecular and immunohistochemical biomarkers correlating with known clinical prognostic factors and outcome.

XII. To evaluate the hepatoblastoma molecular risk-predictive model (HB-MRP) to risk stratify hepatoblastoma patients in the context of the current AHEP1531 trial.

XIII. To collect for future analysis samples to assess the pharmacogenomics (PG) related to cisplatin therapy in pediatric and adolescent liver tumor patients and correlate PG with Boston Grading Scale for ototoxicity.

XIV. To collect for future analysis samples such that novel biomarkers of renal toxicity (urine neutrophil gelatinase-associated lipocalin [NGAL], cystatin C and Kim1) from cisplatin therapy can be correlated with pharmacogenomics, other associated toxicities, and outcomes.

XV. To determine which system (Children's Oncology Group [COG] PRETEXT, SIOPEL PRETEXT, or a new hybrid definition of PRETEXT) of the annotation factors for V, P, E, F and R provides the best prognostic information for determining response to chemotherapy, guiding risk based therapy, predicting surgical resectability, and EFS.

XVI. To determine the concordance between institutional and expert panel review assessment of PRETEXT and POSTTEXT stage in an international cooperative group setting.

OUTLINE:

GROUP A (VERY LOW RISK HB): Patients are assigned to 1 of 2 groups.

GROUP A1 (WDF): Patients undergo observation.

GROUP A2 (NON-WDF): Patients receive cisplatin (CDDP) intravenously (IV) over 6 hours on day 1 following surgery. Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

GROUP B (LOW RISK HB): Patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 14 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients are then assigned to 1 of 2 groups.

GROUP B1 (RESECTABLE): Patients receive 2 cycles of cisplatin, undergo surgery, then are randomized to 1 of 2 arms (2 vs 4 additional cycles of cisplatin).

GROUP B1 ARM 4-CDDP: Patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 14 days for up to 4 total cycles (2 pre-surgery, 2 post-surgery) in the absence of disease progression or unacceptable toxicity.

GROUP B1 ARM 6-CDDP: Patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 14 days for up to 6 total cycles (2 pre-surgery, 4 post-surgery) in the absence of disease progression or unacceptable toxicity.

GROUP B2 (UNRESECTABLE): Patients receive 2 cycles of cisplatin, then are assigned to 1 of 2 arms (resectable vs unresectable).

GROUP B2 ARM I (RESECTABLE): Patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 14 days for up to 6 total cycles (4 pre-surgery, 2 post-surgery). After cycle 4, patients undergo surgery, then continue with 2 additional cycles of cisplatin.

GROUP B2 ARM II (UNRESECTABLE): Patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 14 days for up to 6 total cycles.

GROUP C (INTERMEDIATE RISK HB): Patients are randomized to 1 of 2 arms.

GROUP C ARM CDDP: Patients receive cisplatin IV over 6 hours on day 1. Treatment repeats every 14 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo surgery after cycle 2 or 4.

GROUP C ARM C5VD: Patients receive cisplatin IV over 6 hours on day 1, 5-fluorouracil IV over 1-15 minutes, vincristine sulfate IV over 1 minute on days 1, 8, and 15 and doxorubicin IV over 1-15 minutes on days 1 and 2. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo surgery after cycle 2 or 4.

GROUP D (HIGH RISK HB): SIOPEL-4 IV INDUCTION: Patients receive cisplatin IV over 6 hours on days 1, 8, and 15 (for cycles 1 and 2) and days 1 and 8 (for cycle 3) and doxorubicin IV over 1-15 minutes on days 8 and 9 (for cycles 1 and 2) and days 1 and 2 (for cycle 3). Cycles 1 and 2 are 28 days; cycle 3 is 21 days. Patients are then assigned to 1 of 2 arms.

GROUP D1: CONSOLIDATION THERAPY: Patients with lung complete remission (either with chemotherapy and/or surgery) receive carboplatin IV over 1 hour on day 1 and doxorubicin IV over 1-15 minutes on days 1 and 2. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity.

GROUP D2: Patients with residual metastatic disease are randomized to 1 of 2 arms.

GROUP D2 ARM CE: Patients receive carboplatin IV over 1 hour on days 1 and 2, doxorubicin IV over 1-15 minutes on days 1 and 2 during cycles 1, 3 and 5, and carboplatin IV over 1 hour and etoposide IV over 2 hours on day 1 and 2 of cycles 2, 4 and 6. Treatments repeat every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

GROUP D2 ARM VI: Patients receive carboplatin IV over 1 hour on days 1 and 2 and doxorubicin IV over 1-15 minutes on days 1 and 2 during cycles 1, 3 and 5. Patients also receive vincristine sulfate IV over 1 minute on days 1 and 8 and irinotecan IV over 60-90 minutes once daily (QD) on days 1 to 5 of cycles 2, 4 and 6. Treatments repeat every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

GROUP E (RESECTED HCC): Patients are assigned to 1 of 2 groups.

GROUP E1: Patients with HCC secondary to underlying hepatic disease undergo observation only.

GROUP E2 (PLADO): Patients with de novo HCC receive cisplatin IV over 6 hours on day 1 and doxorubicin IV over 1-15 minutes on days 1 and 2 following surgery. Treatments repeat every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

GROUP F (UNRESECTED AND/OR METASTATIC HCC): Patients are randomized to 1 of 2 arms.

GROUP F ARM 1 (PLADO): Patients receive cisplatin IV over 6 hours on day 1, doxorubicin IV over 1-15 minutes on days 1 and 2 and sorafenib orally (PO) twice daily (BID) on days 3-21. Treatments repeat every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients may undergo surgery, if tumors are resectable, or receive an additional 3 cycles of the treatment.

GROUP F ARM 2 (P/GEMOX): Patients receive cisplatin IV over 6 hours on day 1, doxorubicin IV over 1-15 minutes on days 1 and 2 and sorafenib PO BID on days 3-14 of cycles 1 and 3. Patients also receive gemcitabine IV over 90 minutes on day 1, oxaliplatin IV over 2 hours on day 1 and sorafenib PO on days 1-14 of cycles 2 and 4. Patients may undergo surgery, if tumors are resectable, or receive an additional 4 cycles of the treatment.

Patients may undergo blood sample collection on study.

After completion of study treatment, patients are followed up for a minimum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients in Group F must have a body surface area (BSA) >= 0.6 m^2
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must be newly diagnosed with histologically-proven primary pediatric hepatic malignancies including hepatoblastoma or hepatocellular carcinoma, except as noted below; patients with a diagnosis of hepatocellular neoplasm, not otherwise specified, should be classified and treated per hepatoblastoma treatment arms; note that rapid central pathology review is required in some cases; please note: all patients with histology as assessed by the institutional pathologist consistent with pure small cell undifferentiated (SCU) HB will be required to have testing for INI1/SMARCB1 by immunohistochemistry (IHC) according to the practices at the institution
* Patients with histology consistent with pure SCU must have positive INI1/SMARCB1 staining
* For all Group A patients, WDF status as determined by rapid review will be used to further stratify patients to Group A1 or A2

  * For Groups B, C and D, rapid review is required if patients are either >= 8 years of age or have an alphafetoprotein (AFP) =< 100 at diagnosis
  * For all Groups E and F patients, rapid central pathology review is required
* In emergency situations when a patient meets all other eligibility criteria and has had baseline required observations, but is too ill to undergo a biopsy safely, the patient may be enrolled without a biopsy

  * Clinical situations in which emergent treatment may be indicated include, but are not limited to, the following circumstances:

    * Anatomic or mechanical compromise of critical organ function by tumor (e.g., respiratory distress/failure, abdominal compartment syndrome, urinary obstruction, etc.)
    * Uncorrectable coagulopathy
  * For a patient to maintain eligibility for AHEP1531 when emergent treatment is given, the following must occur:

    * The patient must have a clinical diagnosis of hepatoblastoma, including an elevated alphafetoprotein (AFP), and must meet all AHEP1531 eligibility criteria at the time of emergent treatment
    * Patient must be enrolled on AHEP1531 prior to initiating protocol therapy; a patient will be ineligible if any chemotherapy is administered prior to AHEP1531 enrollment
  * Note: If the patient receives AHEP1531 chemotherapy emergently PRIOR to undergoing a diagnostic biopsy, pathologic review of material obtained in the future during either biopsy or surgical resection must either confirm the diagnosis of hepatoblastoma or not reveal another pathological diagnosis to be included in the analysis of the study aims
* Patients may have had surgical resection of the hepatic malignancy prior to enrollment; all other anti-cancer therapy for the current liver lesion is prohibited
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 or

  * A serum creatinine based on age/gender as follows:

    * Age: maximum serum creatinine (mg/dL)
    * 1 month to < 6 months: 0.4 (male and female)
    * 6 months to < 1 year: 0.5 (male and female)
    * 1 to < 2 years: 06 (male and female)
    * 2 to < 6 years: 0.8 (male and female)
    * 6 to < 10 years: 1 (male and female)
    * 10 to < 13 years: 1.2 (male and female)
    * 13 to < 16 years: 1.5 (male), 1.4 (female)
    * >= 16 years: 1.7 (male), 1.4 (female)
* Total bilirubin =< 5 x upper limit of normal (ULN) for age
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 10 x upper limit of normal (ULN) for age
* Shortening fraction of >= 28% by echocardiogram (for patients on doxorubicin-containing regimens [Groups C, D, E2, and F] assessed within 8 weeks prior to study enrollment) or
* Ejection fraction of >= 47% by echocardiogram or radionuclide angiogram (for patients on doxorubicin-containing regimens [Groups C, D, E2, and F] assessed within 8 weeks prior to study enrollment)
* Group F patients only: QT/corrected QT (QTc) interval =< 450 milliseconds for males and =< 470 milliseconds for females (assessed within 8 weeks prior to study enrollment)
* Normal pulmonary function tests (including diffusion capacity of the lung for carbon monoxide [DLCO]) if there is clinical indication for determination (e.g. dyspnea at rest, known requirement for supplemental oxygen) (for patients receiving chemotherapy [Groups A, B, C, D, E2, F]); for patients who do not have respiratory symptoms or requirement for supplemental oxygen, pulmonary function tests (PFTs) are NOT required
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Prior chemotherapy or tumor directed therapy (i.e. radiation therapy, biologic agents, local therapy (embolization, radiofrequency ablation, and laser); therefore, patients with a pre-disposition syndrome who have a prior malignancy are not eligible
* Patients who are currently receiving another investigational drug
* Patients who are currently receiving other anticancer agents
* Patients with uncontrolled infection
* Patients who previously received a solid organ transplant, other than those who previously received an orthotopic liver transplantation (OLT) as primary treatment of their hepatocellular carcinoma
* Patients with hypersensitivity to any drugs on their expected treatment arm
* Group C: Patients who have known deficiency of dihydropyrimidine dehydrogenase (DPD)
* Group D:

  * Patients with chronic inflammatory bowel disease and/or bowel obstruction
  * Patients with concomitant use of St. John's wort, which cannot be stopped prior to the start of trial treatment
* Group F:

  * Patients with peripheral sensitive neuropathy with functional impairment
  * Patients with a personal or family history of congenital long QT syndrome
* These criteria apply ONLY to patients who may receive chemotherapy (all groups other than Group E1):

  * Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs; a pregnancy test is required for female patients of childbearing potential
  * Lactating females who plan to breastfeed their infants
  * Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation

    * Note for Group F: patients of childbearing potential should use effective birth control during treatment with sorafenib and for at least 2 weeks after stopping treatment

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 537 (Estimated)
Dates: Start 2018-05-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 3 years
  EFS is defined as the time from randomization (or registration into the trial for non-randomized patients) to the first failure event where the failure events are defined as: progression of existing disease or occurrence of disease at new sites, death from any cause prior to disease progression, or diagnosis of a second malignant neoplasm. Patients who have not had an event will be censored at their last follow-up date. EFS for group A, group B1, group C, group D1, group D2 and E will be presented.
Percentage of Group B2 participants with resectable tumors | 6 months
  Group B patients who are unresectable after cycles 1 & 2 of cisplatin treatment will be assigned to Group B2. These patients will receive cycles 3-6 of cisplatin treatment.
Response rate for Group F patients | Up to 5 years
  Response is defined as complete (CR) or partial (PR) response according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria. Patients who are not assessable for response - e.g. because of early stopping of treatment or death - will be classified as non-responders.

OTHER OUTCOMES:
Failure free survival | 3 years
  Failure free survival is defined as the time from randomization (or registration into the trial for non-randomized patients) to first failure event. Failure events are: progression of existing disease or occurrence of disease at new sites, death from any cause prior to disease progression, diagnosis of a second malignant neoplasm, or failure to go to resection.
Overall survival | 3 years
  Overall survival is defined as the time from randomization (or registration for non-randomized patients) to death from any cause.
Percentage of patients experiencing grade 3 or higher adverse events | 8 months
  The percentage of patients experiencing grade 3 or higher toxicity will be reported, where adverse events are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Percentage of patients with chemotherapy-related cardiac, nephro- and oto-toxicity | Up to 5 years
  Adverse events are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Percentage of patients with hearing loss | Up to 5 years
  Hearing loss will be measured according to the SIOP Boston Scale for ototoxicity.
Best response | Up to 5 years
  Response in hepatocellular carcinoma (HCC) will be defined as complete (CR) or partial (PR) response according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria. Response in HB will be defined as CR or PR based on radiological response (RECIST v1.1) and AFP decline.
Percentage of participants who are surgically resectable | Up to 5 years
  Surgical resectability is defined as complete resection, partial resection or transplant following randomization (or enrollment for non-randomized patients).
Percentage of participants with adherence to surgical guidelines | Up to 5 years
  Adherence to surgical guidelines is defined as the local clinician's surgical decision to resect or not compared to the current SIOPEL surgical guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Tiao, Principal Investigator — Children's Oncology Group
Locations (205):
- United States (180):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (13):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia